CLINICAL TRIAL: NCT03735394
Title: Labial Gingival and Osseous Thickness of Upper and Lower Incisors in Thick and Thin Biotypes
Brief Title: Ultrasonic vs Radiographic Measurement of Gingival Biotype. A Novel Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Juan Rossell, assitant professor. Doctor in medical science, Universitat Internacional de Catalunya
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ORT-ECL-2013-03
Record Dates: First submitted 2018-10-13; First posted 2018-11-08 (Actual); Last update posted 2018-11-08 (Actual); Status verified 2018-11

CONDITIONS: Gingival Recession
Keywords: Gingival thickness; gingival biotype; gingival recession; maxilla; mandible
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gingival Biotype (Experimental): A Periodontal probe was used to differentiate between thick and thin biotypes and patients were classified into 3 possible categories of Gingival Biotype (A1, A2 and B) according to Müller & Eger (https://doi.org/10.1034/j.1600-051x.2000.027009621.x). On each group two measurements were taken on the most protruded lower and upper central incisor: 1/ a tangential radiographic film and 2/ an ultrasonic probe measurement with the PIROP Biometric scanner (G-scan) form Echoson
  Interventions: Diagnostic Test: ultrasonic probe

INTERVENTIONS:
Diagnostic Test: ultrasonic probe — apply the head of the ultrasonic probe on the keratinized tissue of the most protruded upper and lower central incisor in order to measure tissue thickness.
  Other Names: tangential x-ray

SUMMARY:
This clinical study consists on taking 2 different records of the upper and lower incisors area : 1) a perpendicular x-ray and 2) an ultrasonic measurement of gingival thickness on the labial plate. Both measurements are used in order to measure gingival and bone thickness.

The aim was to verify the reliability of the tissue measurements of an ultrasonic technique compared with the radiographic technique and to verify whether the biotype has correlation between the maxillary and mandibular biotype in the same patient.

DETAILED DESCRIPTION:
The examination of the patients included:

* One color photograph of the upper and lower incisors complex with the periodontal probe introduced on the gingival sulcus
* Gingival thickness of the most protruded upper and lower incisors was measured with the biometric scanner PIROP. A lip expander was placed and clorhexidine gel was applied on top of the ultrasonic head for better wave conduction. Measurements were taken 10 times at the same point and a mean measurement was obtained.
* A tangential radiograph was taken on each patient perpendicular to the axis of the crown of the central upper and lower incisors with a periapical film holding system, and a metal strip (5mm x 1mm x 0,1mm) placed labial to the keratinized gingiva following the inclination of the incisor. A lip expander was used to keep the lips from touching the metal strip. Air was blown over the attached gingiva before placing the metal strip. The metal strip was placed along the long axis of the most protruded lower incisor crown.

All patients were evaluated and categorized in one of three possible categories: A1 (7 patients, 23,3%), A2 (12 patients, 40%), and B (11 patients, 36,7%). The patients were assigned into each category by two examiners, according to the visual and clinical aspect of the keratinized gingiva in the lower incisors. Group A1 and A2 both had thin keratinized gingiva and differed in width (group A1 comprised values ≤2mm, and group A2 had width values >2mm of keratinized gingiva). Group B comprised thick and wide keratinized gingiva. Width of gingiva was measured with a periodontal probe. Thickness of gingiva was assessed by probe transparency, where the examiner determined whether the periodontal probe was visible through the marginal soft tissue.

Radiographic measurements

Radiographs were scanned at a 1:1 scale. Scanned images were saved in JPEG format. Millimetric measurements were made using the Adobe Photoshop program to a 0.1mm precision. Four measurements were taken on each radiograph:

1. Gingival thickness on the upper incisor
2. Bone thickness on the upper incisor
3. Gingival thickness on the lower incisor
4. Bone thickness on the lower incisor

Gingival thickness was measured on the radiographs to compare it with the measurements taken with the biometric scanner. This was a founded and a reliable method to validate the use of the scanner. A master file was created and the data were statistically analyzed using a statistical software package.

Size of the sample was obtained with the correlation of lower gingiva and thickness of lower gingiva. The result was 26 calculated with the correlation coefficient 0,587. A 20% tax of follow-up loss was estimated.

Intraexaminer reliability was determined using intraclass correlation coefficient (ICC) with a positive confidence interval at 95% (IC 95%). An ICC was used to compare the valid method for group classification between visual and probe transparency methods.

The data were subjected to 95% confidence interval for the mean of all variables. The strength of correlation was determined by a P value <0.05, which was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or older,
* presence of all lower incisors
* good periodontal health without bone loss or gingival inflammation
* no dental compensations of skeletal malocclusion
* crowding of less than 4mm
* no history of dental or traumatic lesions in lower incisors

Exclusion Criteria:

* gingival inflammation
* daily smokers
* patients taking drugs that causes gingival inflammation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-04-15 (Actual); Primary Completion 2017-05-22 (Actual); Study Completion 2017-09-08 (Actual)

PRIMARY OUTCOMES:
compare between maxilla and mandibular biotype measured with the periodontal probe | 1 day
  Classify all patients into one of the three established categories (A1, A2, B) with the aid of a periodontal probe, and compare within the same patient if the biotype of maxilla and mandible is the same or it differs

SECONDARY OUTCOMES:
Differences in tissue thickness according to gender | 1 day
  Classify patients in male or female and measure tissue thickness regardless of the biotype measured with both the radiographic technique and ultrasonic device
thickness biotype differences | 1 day
  establish a possible correlation between maxilla and mandible tissue thickness according to the three possible established categories of biotype measured with radiographic technique and ultrasonic device

CONTACTS AND LOCATIONS:
Overall Officials: Andreu Puigdollers, Study Director — Chairman
Locations (1):
- Universitat Internacional de Catalunya, Sant Cugat del Vallès, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
All identified data of individuals measurements will be available
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: data will be available during 1 year of study completion
Access Criteria: Data access requests will be reviewed by an external reviewer, if any requestor wants access there will be a need to sign a data access agreement

REFERENCES:
- [Background] Eghbali A, De Rouck T, De Bruyn H, Cosyn J. The gingival biotype assessed by experienced and inexperienced clinicians. J Clin Periodontol. 2009 Nov;36(11):958-63. doi: 10.1111/j.1600-051X.2009.01479.x. Epub 2009 Oct 6. PMID 19811580
- [Background] Zweers J, Thomas RZ, Slot DE, Weisgold AS, Van der Weijden FG. Characteristics of periodontal biotype, its dimensions, associations and prevalence: a systematic review. J Clin Periodontol. 2014 Oct;41(10):958-71. doi: 10.1111/jcpe.12275. Epub 2014 Aug 27. PMID 24836578